CLINICAL TRIAL: NCT05094921
Title: Effect of Hydrotherapy (Halliwick Concept)on Motor Function in Spastic Cerebral Palsy: A Randomized Controlled Trial
Brief Title: Halliwick Concept on Motor Functions in Spastic CP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: October 6 University (Other)
Responsible Party: Principal Investigator, Mohamed Magdy Ali Hassan ElMeligie, Principal investigator, October 6 University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Halliwick07
Record Dates: First submitted 2021-09-17; First posted 2021-10-26 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Spastic Cerebral Palsy; Spastic Hemiplegic Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Halliwick method group) (Experimental): Under water exercise program according to halliwick concept which will be applied as three sessions per week for three successive months. Underwater exercises will be performed under the supervision of a certified aquatic therapist. This practitioner will instruct the child in proper techniques for performing exercises while ensuring child's safety by using flotation devices, body boards or float belts when necessary. Also the pool where the children will perform underwater exercises will be equipped with ramps, chair lifts, stairs, and handrails to facilitate a child's ability to access the pool.
  Interventions: Other: Aquatic Halliwick method
- Group B (conventional physical therapy group) (Active Comparator): Conventional selected exercise program for 60 minutes , three sessions per week for three successive months aiming to improve the motor functions of the children in form of: (1) Neuro-developmental technique, (2) Back and abdominal exercises, (3) improving postural responses, (4) Flexibility exercises, (5) Strengthening exercise (particularly knee extensors, hip abductors and the ankle dorsi-flexors muscles) and (6) Improving standing, weight transfer and shift and finally facilitation of normal walking pattern .
  Interventions: Procedure: Conventional physical therapy

INTERVENTIONS:
Other: Aquatic Halliwick method — The Halliwick Concept is a detailed swimming programme based on the scientific principles of body mechanics and the properties of water intended to educate individuals with special needs to be water safe and to move independently in the water as much as possible (Lambeck & Stanat 2001a).The programme consists of 10 specific progressive stages that are achieved without the use of floatation devices (Lambeck & Stanat 2001b).
  Arms: Group A (Halliwick method group)
Procedure: Conventional physical therapy — Conventional selected exercise program for 60 minutes ,3 session per week for 3 successive months aiming to improve the motor functions of the children in form of: (1) Neuro-developmental technique, (2) Back and abdominal exercises to improve postural control and correct spinal deformities (3) improving postural responses, (4) Flexibility exercises of the soft tissue (5) Strengthening exercise (particularly knee extensors, hip abductors and the ankle dorsi-flexors muscles and (6) Improving standing, weight transfer and shift and finally facilitation of normal walking pattern .
  Arms: Group B (conventional physical therapy group)

SUMMARY:
This randomized controlled trial will investigate the effect of hydrotherapy (halliwick concept) on motor functions in children with spastic cerebral palsy (CP). Minimum of 30 Spastic CP children will be recruited for this study. Children will be randomly assigned into control group who will receive conventional selected exercise treatment or study group who will receive the same conventional program in addition to underwater exercise program. Motor function will be evaluated at baseline and after 3 months of treatment. No potential harms are expected during this study.

ELIGIBILITY:
Inclusion Criteria:

* Children from both sexes diagnosed with spastic CP according to a pediatrician
* The degree of spasticity will be determined as grade two or less according to modified Ashworth scale
* Their age will range from five to nine years
* Intelligence quotient score > 35 (no worse than moderate intellectual disability) as assessed via Wechsler test scales
* No severe psychosocial or behavioral problems, such high aggression or risk of self-harm.

Exclusion Criteria:

* Initiation of oral antispastic medication
* botulinum toxin injections or surgery performed less than 90 days before enrollment
* severe visual or auditory impairment
* uncontrollable epilepsy (defined as the occurrence of seizures despite the use of at least one antiepileptic drug)
* open wounds
* children with a psychiatric disorder
* cognitive disorders evaluated by the pediatric evaluation of disability inventory
* uncontrolled epilepsy
* active infection
* severe cardiopulmonary disorders.

Ages: 5 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-09-08 (Actual); Study Completion 2021-09-08 (Actual)

PRIMARY OUTCOMES:
Change from Gross motor function measure at 3 months [ Time Frame: 3 months ] | Baseline and after 3 months
  The Gross Motor Function Measure (GMFM) is an observational clinical tool designed to evaluate change in gross motor function in children with cerebral palsy. There are two versions of the GMFM - the original 88-item measure (GMFM-88) and the more recent 66-item GMFM (GMFM-66) The scoring system of the GMFM is a four-point scale divided into five categories (lying and rolling; sitting; crawling and kneeling; standing; walking, running).

CONTACTS AND LOCATIONS:
Locations (1):
- October 6 University Hospital, Al Ḩayy Ath Thāmin, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
all of the individual participant data collected during the trial and after deidentification
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 6 Months after study publication
Access Criteria: Email: mohamed.magdy.pt@o6u.edu.eg